CLINICAL TRIAL: NCT00726999
Title: Perioperative Use of Gabapentin To Decrease Opioid Requirements in Pediatric Spinal Fusion Patients
Brief Title: Perioperative Use of Gabapentin To Decrease Narcotic Requirements in Spinal Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Lynn Rusy, Professor of Anesthesiology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06/71,GC 138
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2010-12-30 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Pain
Keywords: Gabapentin; Pediatric Spinal Fusion; Narcotic Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Gabapentin
  Interventions: Drug: Gabapentin; Drug: Morphine
- 2 (Placebo Comparator): Placebo Comparator -- pill matched in appearance to gabapentin
  Interventions: Drug: Placebo; Drug: Morphine

INTERVENTIONS:
Drug: Gabapentin — oral gabapentin in load pre-op (15mg/kg) and maintenance 5mg/kg TID for 5 days or discharge
  Other Names: Neurontin
  Arms: 1
Drug: Placebo
  Arms: 2
Drug: Morphine — Administered as needed

SUMMARY:
Blinded study using oral gabapentin in load pre-operative (15mg/kg) and maintenance 5mg/kg three times a day (TID) for 5 days or discharge, Patient Controlled Analgesia (PCA) morphine and placebo group with similar pills, also PCA morphine. The goal is to measure morphine usage and incidence of morphine side effects (pruritis, days foley, days to first stool, sedation, pain scores, PCA use).

DETAILED DESCRIPTION:
Healthy, American Society of Anesthesia (ASA) 1-2 Idiopathic Scoliosis patients for spinal fusion.

Blinded, drug only known by hospital pharmacist. Study group 1- Gabapentin 15mg/kg with premed, 5/kg TID for 5 days of discharge, standard PCA morphine with dose and basal Study Group 2- Capsules resembling neurontin, with standard PCA morphine

No remifentanil, clonidine, ketamine

N=60 First patient enrolled 6/06 Last patient enrolled 7/15/08

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2, Idiopathic Scoliosis

Exclusion Criteria:

* ASA 3 or greater
* Neuromuscular scoliosis
* On narcotics baseline

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2006-06; Primary Completion 2008-07 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn M Rusy, MD, Principal Investigator — Medical College of Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin/Morphine: Gabapentin - group received gabapentin 3 times daily 5 mg/kg/dose. *Both groups received Morphine as needed.
- Placebo/Morphine: Placebo Comparator - group received placebo 3 times daily. *Both groups received Morphine as needed.
Period: Overall Study
Arm/Group | Gabapentin/Morphine | Placebo/Morphine
Started | 32 | 31
Completed | 29 | 30
Not Completed | 3 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin/Morphine | Placebo/Morphine | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 31 | 63
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (2.1) | 14.2 (1.8) | 14.5 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Amount of Morphine Consumed (mg/kg/hr)
Description: Patients are taken to the PARU immediately after surgery, and typically remain for a period of 1 hour.
Time Frame: PARU (Postanesthesia Recovery Unit - participants typically remain in PARU for 1 hour)
Measure: Mean (Standard Deviation); unit: mg/kg/h
Arm/Group | Gabapentin/Morphine | Placebo/Morphine
Number analyzed (Participants) | 32 | 31
mg/kg/h | 0.064 (0.031) | 0.044 (0.017)

2. Primary Outcome: Amount of Morphine Consumed (mg/kg/hr)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mg/kg/h
Arm/Group | Gabapentin/Morphine | Placebo/Morphine
Number analyzed (Participants) | 29 | 30
mg/kg/h | 0.055 (0.017) | 0.046 (0.016)

3. Primary Outcome: Amount of Morphine Consumed (mg/kg/hr)
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: mg/kg/h
Arm/Group | Gabapentin/Morphine | Placebo/Morphine
Number analyzed (Participants) | 29 | 30
mg/kg/h | 0.047 (0.019) | 0.036 (0.016)

4. Secondary Outcome: Number of Ondansetron Doses Administered for Nausea
Description: The number of doses of Ondansetron given for nausea to participants in both groups.
Time Frame: First 10 days after surgery
Measure: Median (Inter-Quartile Range); unit: doses of medication administered
Groups:
- Gabapentin Group: Gabapentin
  Gabapentin: oral gabapentin in load pre-op (15mg/kg) and maintenance 5mg/kg TID for 5 days or discharge
  Morphine: Administered as needed
- Placebo Group: Placebo Comparator -- pill matched in appearance to gabapentin
  Placebo
  Morphine: Administered as needed
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 29 | 30
doses of medication administered | 2.0 [0.0 to 6.0] | 2.0 [0.0 to 3.75]

ADVERSE EVENTS:
Arm/Group | Gabapentin/Morphine | Placebo/Morphine
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes